CLINICAL TRIAL: NCT02770599
Title: IMPROVING THE HEALTH CARE IN INFLAMMATORY BOWEL DISEASE. A Clinical Study Comparing Two Different Outpatient Follow-up Models by Measuring Patient Reported Health Related Quality of Life, Quality of Care, Adherence and Clinical Outcomes.
Brief Title: Improving the Health Care in Inflammatory Bowel Disease.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital of North Norway (Other)
Collaborators: University of Tromso (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/1397(REK)
Record Dates: First submitted 2016-04-04; First posted 2016-05-12 (Estimated); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Crohn Disease; Colitis, Ulcerative
Keywords: IBD; HRQoL; QoC; Adherence; IBD nurse; MDT
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IBD multidisciplinary team model (MDT): IBD multidisciplinary team model including IBD nurse
  Interventions: Other: IBD multidisciplinary team model including IBD nurse
- IBD conventionally follow up model (CF): IBD patient treated by doctors with specialist qualifications, assistant doctors, general practitioner or scarcity of follow-up-service.

INTERVENTIONS:
Other: IBD multidisciplinary team model including IBD nurse — IBD multidisciplinary team model including IBD nurse
  Groups: IBD multidisciplinary team model (MDT)

SUMMARY:
Inflammatory Bowel Disease (IBD) refers to two chronic diseases (Crohn's disease and Ulcerative colitis) both complex disorders requiring a long-term management, with significant healthcare resource consumption. Traditionally IBD patients has been treated by a variety of health care professional including doctors with specialist qualifications, assistant doctors, general practitioner or scarcity of follow-up-service. Lately there has been a shift in the health care service from conventional follow - up (CF) to a rising numbers of health care models in term of Multidisciplinary team (MDT) also including care for IBD patients. MDT- models have been identified as important for continuity in patient centred care where nurses have a key role within the team by enhancing patient care. Patients have directly access to the IBD nurse who performing independently consultations at the IBD - Policlinic. This study will test the hypothesis that MDT including an IBD - nurse is preferable concerning; patient reported Health Related Quality of Life (HRQoL) Quality of Care (QoC), and clinical outcomes including adherence. This will be a retrospective clinical quality survey with a single time point measurement, with consecutive recruitments of patients in the course of a 12-month period. Data will be collected from medical records and patient questionnaires. Investigators plan involving 300 participants aged >18 and < 80 recruited from Medical departments in North Norway and from Diakonhjemmet in Oslo. Half will be from CF-models and half from the IBD - MDT. The study have approval from the local Ethics committee and application to the Data protection Officer has been submitted. All participants are asked for provide written consent. The results can potentially contribute; to a better utilization of health care resources, improve quality of health and quality of care. In a nurse-perspective, this organising model can be valuable in recruiting nurses by presenting a new challenging task concept, and identify the gaps in their own knowledge and skills. A well-established MDT can also be reasonable in a cost effective way by decreasing hospitalisation and fee up clinical spaces for the gastroenterologist.

ELIGIBILITY:
Inclusion Criteria:

* Diagnose duration > 2 years, to ensure that the patients have some experience with IBD and their follow-up system, respectively

Exclusion Criteria:

* Non-Norwegian patients who will have difficulties understanding the questionnaires
* patients with cognitive disabilities

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Inflammatory bowel disease belonging two different out patient follow-up models; IBD multidisciplinary team including IBD specialist nurse or conventionally follow -up model, respectively.
Sampling Method: Non-Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2016-05-15 (Actual); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life | during autumn of 2016
  Health Related Quality of Life measured by The inflammatory Bowel Disease Questionnaire (IBDQ). This is a disease specific valid, reliable and sensitive instrument for clinical trials designed to measure the effects of the IBD on daily function and quality of life during the past two weeks. An absolute change on 16 of 224 points in total score has been used to define a minimum clinically important difference.

SECONDARY OUTCOMES:
Quality of care | during autumn of 2016
  The questionnaire QUOTE IBD focus on GP-care and medical specialist care. This is a short, valid and reliable questionnaire. The answers is divided into four categories: "not important" - fairly important - important - extremely important" and " no - not really - on the whole yes - yes".

OTHER OUTCOMES:
Adherence associated to IBD medications | during autumn of 2016
  The questionnaire Morisky Medication Adherence Scale (MMAS) is a validated 8-question measuring scale for medication adherence in IBD patients. The patients can score from 0-8 points, where score > 2 = low adherence and a score of 1 or 2 = medium adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Ragnhild Broderstad, Ph.D, Principal Investigator — The Health Faculty, Institute of Community Health,
Locations (1):
- University Hospital of North Norway, Harstad, Norway

IPD SHARING:
Plan to Share IPD: No